CLINICAL TRIAL: NCT01577550
Title: Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of Single Rising i.v. (Stage 1) and s.c. (Stage 2) Doses of BI 655066 in Male and Female Patients With Moderate to Severe Psoriasis (Randomised, Double-blind, Placebo-controlled Within Dose Groups)
Brief Title: Single Rising Dose Study of BI 655066 in Patients With Moderate and Severe Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1311.1; 2012-000081-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-04-10; First posted 2012-04-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Psoriasis
Keywords: ABBV-066; BI 655066; risankizumab
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

ARMS (4):
- i.v. BI 655066 (Experimental): A subject to receive a single i.v. dose of BI 655066
  Interventions: Drug: BI 655066 (very high i.v. dose); Drug: BI 655066 (low i.v. dose); Drug: BI 655066 (high medium i.v. dose); Drug: BI 655066 (very low i.v. dose); Drug: BI 655066 (high i.v. dose); Drug: BI 655066 (low medium i.v. dose)
- i.v. placebo (Placebo Comparator): A subject to receive a single i.v. dose of placebo
  Interventions: Drug: Placebo, i.v.
- s.c. BI 655066 (Experimental): A subject to receive a single s.c. dose of BI 655066
  Interventions: Drug: BI 655066 (high s.c. dose); Drug: BI 655066 (low s.c. dose)
- s.c. placebo (Placebo Comparator): A subject to receive a single s.c. dose of placebo
  Interventions: Drug: Placebo, s.c.

INTERVENTIONS:
Drug: BI 655066 (very high i.v. dose) — Single very high i.v. dose BI 655066
  Other Names: ABBV-066; risankizumab
  Arms: i.v. BI 655066
Drug: Placebo, i.v. — Single i.v. administration of placebo
  Arms: i.v. placebo
Drug: BI 655066 (high s.c. dose) — Single high s.c. dose BI 655066
  Other Names: ABBV-066; risankizumab
  Arms: s.c. BI 655066
Drug: BI 655066 (low i.v. dose) — Single low i.v. dose BI 655066
  Other Names: ABBV-066; risankizumab
  Arms: i.v. BI 655066
Drug: BI 655066 (high medium i.v. dose) — Single high medium i.v. dose BI 655066
  Other Names: ABBV-066; risankizumab
  Arms: i.v. BI 655066
Drug: BI 655066 (very low i.v. dose) — Single very low i.v. dose BI 655066
  Other Names: ABBV-066; risankizumab
  Arms: i.v. BI 655066
Drug: BI 655066 (low s.c. dose) — Single low s.c. dose BI 655066
  Other Names: ABBV-066; risankizumab
  Arms: s.c. BI 655066
Drug: BI 655066 (high i.v. dose) — Single high i.v. dose BI 655066
  Other Names: ABBV-066; risankizumab
  Arms: i.v. BI 655066
Drug: Placebo, s.c. — Single s.c. administration of placebo
  Other Names: ABBV-066; risankizumab
  Arms: s.c. placebo
Drug: BI 655066 (low medium i.v. dose) — Single low medium i.v. dose BI 655066
  Other Names: ABBV-066; risankizumab
  Arms: i.v. BI 655066

SUMMARY:
Safety, tolerability and efficacy of BI 655066 in male and female patients with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients aged 18-75 years (inclusive)
2. Chronic moderate to severe plaque psoriasis lasting =>6 months with involvement of Body Surface Area (BSA) =>10%, Psoriasis Area and Severity Index (PASI) =>12 and Static Physician Global Assessment (sPGA) score of moderate and above
3. Body Mass Index (BMI) =>18.5 and <40 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation
5. Female patients must not be of childbearing potential (i.e., must be postmenopausal or surgically sterilized) and must have a negative pregnancy test at screening.

Exclusion criteria:

1. Evidence of current or previous clinically significant disease, medical condition other than psoriasis, or finding of the medical examination (including vital signs and Electrocardiogram (ECG)), that in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data. This criterion provides an opportunity for the investigator to exclude patients based on clinical judgment, even if other eligibility criteria are satisfied (Psoriatic arthritis is not considered an exclusion.)
2. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders, chronic or relevant acute infections including hepatitis and tuberculosis (or a positive interferon-gamma release assay at screening) or history of orthostatic hypotension, fainting spells or blackouts, that in the investigator's judgement, could jeopardize the safe conduct of the study
3. History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients
4. Use of biologic agents or psoralen and ultraviolet A (PUVA) within 12 weeks prior to Visit 2, ultraviolet B (UVB) phototherapy and oral anti-psoriatic medications within 4 weeks prior to Visit 2, or topical anti-psoriasis medications (except emollients) within 2 weeks prior to Visit 2
5. Use of ustekinumab within 24 weeks prior to Visit 2
6. Had a prior treatment of psoriasis with biologics with inadequate clinical response to therapy as assessed by a dermatologist or the investigator
7. Intake of restricted medications or drugs considered likely to interfere with the safe conduct of the study
8. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval within 10 days prior to administration or during the trial
9. Participation in another trial with an investigational drug within 4 weeks or 5 half-lives (whichever is greater) preceding Visit 2
10. History of alcohol abuse within last 12 months (intake of more than 30 g/day)
11. History of drug abuse within last 12 months or positive drug screen at screening or Visit 2
12. Any blood donation or significant blood loss within 4 weeks prior to Visit 2
13. Unwilling or not capable to abstain from alcoholic beverages one day prior and two days after Visit 2
14. Excessive physical activities (within 1 week prior to Visit 2)
15. Any laboratory value at the screening visit outside the reference range that is of clinical relevance based on physician investigator judgement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with good and satisfactory assessment of global tolerability by investigator | 24 weeks
Number of patients without any symptoms at the drug administration site, at per local assessment of tolerability by investigator | up to 1 week
Number of participants with adverse events | up to 24 weeks
Number of participants with clinically relevant findings in vital signs | up to 24 weeks
Number of participants with clinically significant abnormalities in electrocardiogramm (ECG) results | up to 24 weeks
Number of participants with significant changes from baseline laboratory measurements | up to 24 weeks

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (absolute score) | up to 24 weeks
Percentage of participants with Static Physicians Global Assessment (clear and almost clear) | up to 24 weeks
Cmax (maximum measured concentration of the analyte in plasma) | up to 24 weeks
tmax (time from dosing to maximum measured concentration) | up to 24 weeks
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | 24 weeks
Psoriasis Area and Severity Index (percentage change from baseline) | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Chair — AbbVie
Locations (9):
- United States (7):
  - 1311.1.0007 Boehringer Ingelheim Investigational Site, Burbank, California
  - 1311.1.0008 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1311.1.0003 Boehringer Ingelheim Investigational Site, Port Orange, Florida
  - 1311.1.0005 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 1311.1.0006 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1311.1.0004 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1311.1.0002 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
- 1311.1.4901 Boehringer Ingelheim Investigational Site, Berlin, Germany
- 1311.1.0009 Boehringer Ingelheim Investigational Site, Leeds, United Kingdom

REFERENCES:
- [Derived] Suleiman AA, Minocha M, Khatri A, Pang Y, Othman AA. Population Pharmacokinetics of Risankizumab in Healthy Volunteers and Subjects with Moderate to Severe Plaque Psoriasis: Integrated Analyses of Phase I-III Clinical Trials. Clin Pharmacokinet. 2019 Oct;58(10):1309-1321. doi: 10.1007/s40262-019-00759-z. PMID 31054118